CLINICAL TRIAL: NCT01560832
Title: Descriptive Epidemiology of Clostridium Difficile Infection in Hospitalized Adult Patients in the Asia Pacific Region
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0382
Record Dates: First submitted 2012-03-02; First posted 2012-03-22 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laboratory (PCR)-confirmed C.difficile infection: patient who has experienced the passage of 3 or more unformed or loose stools [diarrhea] conforming to the shape of a container within a 24-hour period and has a positive laboratory test result confirmed by PCR.

SUMMARY:
Clostridium difficile is an important pathogen, causing disease that ranges from mild self-limited diarrhea to life-threatening pseudomembranous colitis. It is estimated that C. difficile is responsible for 10% to 25% of all cases of antibiotic-associated diarrhea and for almost all cases of pseudomembranous colitis. C. difficile disease is mediated by two large toxins, A and B. The toxins damage intestinal epithelial cells and cause the clinical illness. Primary risk factors for C. difficile clinically apparent infection include antimicrobial therapy, hospitalization, residence in a long-term care facility, older age (≥ 65 years), and increased length of hospital stay. The incidence of CDI both in the hospital and the community is important in the understanding and characterization of the disease and its prevention. This observational, epidemiological study will advance the investigators understanding of CDI risk factors in several hospitals and possibly the community in the Asia Pacific region.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged ≥ 20 years at the time of hospitalization in specified wards
* PCR-diagnosed CDI while at the hospital
* Informed consent has been obtained from patients as required by local requirements

Exclusion Criteria:

* Age < 20 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who has experienced the passage of 3 or more unformed or loose stools [diarrhea] conforming to the shape of a container within a 24-hour period and has a positive laboratory test result confirmed by PCR.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To estimate the incidence of laboratory-confirmed hospital-onset CDI cases for hospitalized adult patients | every 5 days after consented to enroll the exam
  A laboratory-confirmed CDI case is defined as a patient who has experienced the passage of 3 or more unformed or loose stools [diarrhea] conforming to the shape of a container within a 24-hour period and has a positive laboratory test result confirmed by PCR. A hospital onset case is defined as a patient with diarrhea more than 48 hours after admission to a hospital.
  The study period is the study duration, which is defined as the first date of surveillance at each hospital until the sample collection date of the last CDI positive patient (N=100).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Gerding DN, Olson MM, Peterson LR, Teasley DG, Gebhard RL, Schwartz ML, Lee JT Jr. Clostridium difficile-associated diarrhea and colitis in adults. A prospective case-controlled epidemiologic study. Arch Intern Med. 1986 Jan;146(1):95-100. PMID 3942469
- [Background] Anand A, Bashey B, Mir T, Glatt AE. Epidemiology, clinical manifestations, and outcome of Clostridium difficile-associated diarrhea. Am J Gastroenterol. 1994 Apr;89(4):519-23. PMID 8147353
- [Background] Bartlett JG. Clostridium difficile: history of its role as an enteric pathogen and the current state of knowledge about the organism. Clin Infect Dis. 1994 May;18 Suppl 4:S265-72. doi: 10.1093/clinids/18.supplement_4.s265. PMID 8086574
- [Background] McDonald LC, Coignard B, Dubberke E, Song X, Horan T, Kutty PK; Ad Hoc Clostridium difficile Surveillance Working Group. Recommendations for surveillance of Clostridium difficile-associated disease. Infect Control Hosp Epidemiol. 2007 Feb;28(2):140-5. doi: 10.1086/511798. Epub 2007 Jan 25. PMID 17265394
- [Background] Zar FA, Bakkanagari SR, Moorthi KM, Davis MB. A comparison of vancomycin and metronidazole for the treatment of Clostridium difficile-associated diarrhea, stratified by disease severity. Clin Infect Dis. 2007 Aug 1;45(3):302-7. doi: 10.1086/519265. Epub 2007 Jun 19. PMID 17599306